CLINICAL TRIAL: NCT00595764
Title: Counseling for Primary Care Office-based Buprenorphine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0504027657; 5R01DA019511 (NIH); NCT00632151 (obsolete NCT alias)
Record Dates: First submitted 2007-10-03; First posted 2008-01-16 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Opiate Dependence
Keywords: Buprenorphine; Buprenorphine/naloxone; Counseling; Primary care
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Physician Management
  Interventions: Behavioral: Manual-guided Physician Management (PM)
- 2 (Experimental): Physician Management plus Cognitive Behavioral Therapy
  Interventions: Behavioral: Physician Management (PM) combined with on-site manual-guided Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Manual-guided Physician Management (PM) — Manual-guided Physician Management (PM) PM, consistent with federal regulations, is designed to reflect usual care by primary care physicians and includes referral to ancillary services.
  Arms: 1
Behavioral: Physician Management (PM) combined with on-site manual-guided Cognitive Behavioral Therapy (CBT) — CBT is provided by skilled psychologists in weekly sessions for the first 12 weeks and focuses on reducing illicit drug use and increasing Buprenorphine adherence.
  Arms: 2

SUMMARY:
The major goal is to determine whether adding cognitive behavioral therapy to physician management will increase the efficacy of buprenorphine/naloxone treatment in an office-based primary care setting.

DETAILED DESCRIPTION:
To evaluate the need for drug counseling aimed at reducing illicit drug use and increasing buprenorphine/naloxone adherence, the proposed study compares manual-guided Physician Management (PM) and PM combined with on-site manual-guided Cognitive Behavioral Therapy (CBT) in a 24 week randomized clinical trial of buprenorphine/naloxone in a heterogeneous population of opioid dependent patients (N=140) in a primary care clinic. PM, consistent with federal regulations, is designed to reflect usual care by primary care physicians and includes referral to ancillary services. CBT will be provided by skilled psychologists in weekly sessions for the first 12 weeks and focuses on reducing illicit drug use and increasing buprenorphine/naloxone adherence. The study will test the hypothesis that that the addition of CBT to PM will lead to decreased illicit drug use, durable effects after counseling has been discontinued, improved buprenorphine/naloxone adherence and will demonstrate incremental cost-effectiveness in patients receiving buprenorphine/naloxone maintenance in primary care. Primary outcome measures include reductions in illicit opioid use and abstinence achievement, as assessed by weekly urine toxicology testing and self report. Secondary outcome measures include retention in treatment, reductions in cocaine use and HIV risk, decreased criminal activity and improved health and employment status. Utilization and costs of services, spillover effects in the PCC, and patient and staff perceptions of benefits and problems associated with primary care agonist maintenance treatment will also be evaluated. The results of this study will help define the role of professional evidence-based drug counseling in expanding access to treatment with buprenorphine/naloxone.

ELIGIBILITY:
Inclusion Criteria:

* opioid dependence

Exclusion Criteria:

* current dependence on alcohol, cocaine, benzodiazepines or sedatives
* current suicide or homicide risk
* current psychotic disorder or untreated major depression
* inability to read or understand English
* life-threatening or unstable medical problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2005-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Fiellin, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - The APT Foundation, Inc. -- Welch Building, New Haven, Connecticut
  - Yale New Haven Hospital Primary Care Center, New Haven, Connecticut

REFERENCES:
- [Result] Fiellin DA, Barry DT, Sullivan LE, Cutter CJ, Moore BA, O'Connor PG, Schottenfeld RS. A randomized trial of cognitive behavioral therapy in primary care-based buprenorphine. Am J Med. 2013 Jan;126(1):74.e11-7. doi: 10.1016/j.amjmed.2012.07.005. PMID 23260506
- [Derived] McHugh RK, Bailey AJ, McConaghy BA, Weiss RD, Fiellin DA, Hillhouse M, Moore BA, Fitzmaurice GM. Behavioral Therapy as an Adjunct to Buprenorphine Treatment for Opioid Use Disorder: A Secondary Analysis of 4 Randomized Clinical Trials. JAMA Netw Open. 2025 Aug 1;8(8):e2528529. doi: 10.1001/jamanetworkopen.2025.28529. PMID 40833692

RESULTS

PARTICIPANT FLOW:
Groups:
- Physician Management: Physician management was provided during fifteen to twenty minute sessions by Internal Medicine physicians with experience providing buprenorphine. Sessions occurred weekly for the first two weeks, every two weeks for the next four weeks, then monthly. During physician management the physician followed a structured note that reviewed the patient's recent drug use, provided brief advice on how to achieve or maintain abstinence, supported efforts to reduce drug use or remain abstinent, reviewed medical and psychiatric complaints, assessed social, work and legal function, discussed weekly urine toxicology results and reviewed attendance at self-help groups.
- Physician Management Plus Cognitive Behavioral Therapy: In addition to recieving Physician Management identical to the Physician Management only condition, patients were offered up to 12, 50-minute weekly sessions during the first 12 weeks of treatment. Cognitive behavioral therapy was provided by masters- and doctoral-level clinicians who were trained to competence using a manual adapted from the use of cognitive behavioral therapy for cocaine dependence. To ensure fidelity, all sessions were audio- or video-taped, and clinicians underwent weekly supervision. The main components of counseling focused on a functional analysis of behavior, behavioral activation, identifying and coping with drug cravings, enhancing drug-refusal skills, enhancing decision making about high-risk situations and improve problem-solving skills.
Period: Overall Study
Arm/Group | Physician Management | Physician Management Plus Cognitive Behavioral Therapy
Started | 71 | 70
Completed | 32 | 27
Not Completed | 39 | 43
Not completed — Protocol Violation | 24 | 19
Not completed — Missed Medication >1 week | 10 | 17
Not completed — Missed 3 PM visits | 1 | 7
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Physician Management Plus Cognitive Behavioral Therapy: In addition to receiving Physician Management identical to the Physician Management only condition, patients were offered up to 12, 50-minute weekly sessions during the first 12 weeks of treatment. Cognitive behavioral therapy was provided by masters- and doctoral-level clinicians who were trained to competence using a manual adapted from the use of cognitive behavioral therapy for cocaine dependence. To ensure fidelity, all sessions were audio- or video-taped, and clinicians underwent weekly supervision. The main components of counseling focused on a functional analysis of behavior, behavioral activation, identifying and coping with drug cravings, enhancing drug-refusal skills, enhancing decision making about high-risk situations and improve problem-solving skills.
- Total: Total of all reporting groups
Arm/Group | Physician Management | Physician Management Plus Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 71 | 70 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 70 | 141
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (10.3) | 32.8 (8.6) | 33.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 53 | 51 | 104
Region of Enrollment [Number; unit: participants]
  United States | 71 | 70 | 141

OUTCOME MEASURES:

1. Primary Outcome: Illicit Opioid Abstinence
Description: number of weeks of abstinence from illicit opioids, as documented by urine toxicology and self-report. Range 0 - 24.
Time Frame: 6 months
Population: Repeated measures analysis of variance was used to evaluate differences between groups in the maximum number of consecutive weeks of opioid abstinence for the first and second 12 weeks of treatment. We coded missing urine specimens as positive for opioids in our analysis, thus all participants provided data.
Measure: Mean (Standard Deviation); unit: Weeks of Abstinence
Arm/Group | Physician Management | Physician Management Plus Cognitive Behavioral Therapy
Number analyzed (Participants) | 71 | 70
Weeks of Abstinence | 10.29 (8.48) | 10.12 (8.07)
Statistical Analysis 1: Comparison: Physician Management vs Physician Management Plus Cognitive Behavioral Therapy; With an effect size of 0.46, a sample size of 140 will provide a power of >.84 with p<.05 to detect overall differences between the two treatments on the primary outcome measures; Test type: Superiority or Other; p = .91, ANOVA; Mean Difference (Final Values) = 0.16, Standard Error of Mean 1.40

2. Secondary Outcome: Treatment Completion
Description: The number of patients who completed the study (did not meet the criteria for protective transfer baseed on drug use, did not miss medication for more than seven days, or did not miss three or more Physician Management sessions) at 24 weeks.
Time Frame: 6 months
Population: All participants who entered treatment were evaluated for treatment completion.
Measure: Number; unit: participants
Arm/Group | Physician Management | Physician Management Plus Cognitive Behavioral Therapy
Number analyzed (Participants) | 71 | 70
participants | 45 | 39

3. Secondary Outcome: Cocaine Abstinence
Description: Total weeks of cocaine abstinence as documented by weekly urine toxicology analysis. Range from 0 to 24.
Time Frame: 6 months
Population: All participants provided one or more urine screens thus data was based on all participants.
Measure: Mean (Standard Deviation); unit: weeks of abstinence
Arm/Group | Physician Management | Physician Management Plus Cognitive Behavioral Therapy
Number analyzed (Participants) | 71 | 70
weeks of abstinence | 12.4 (7.7) | 13.8 (7.9)
Statistical Analysis 1: Comparison: Physician Management vs Physician Management Plus Cognitive Behavioral Therapy; Test type: Superiority or Other; p = .29, t-test, 2 sided; Mean Difference (Final Values) = 1.40, Standard Error of Mean 1.32

4. Secondary Outcome: Criminal Activity- Addiction Severity Index (ASI) Legal Composite Score.
Description: The ASI Legal Composite score ranges from 0 to 1 with higher scores corresponding to greater legal problems.
Time Frame: 6 months
Population: All participants who completed one or more ASI assessments were included in the analysis.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Physician Management | Physician Management Plus Cognitive Behavioral Therapy
Number analyzed (Participants) | 67 | 64
Scores on a scale | .044 (.011) | .066 (.010)
Statistical Analysis 1: Comparison: Physician Management vs Physician Management Plus Cognitive Behavioral Therapy; Test type: Superiority or Other; p = .58, Mixed Models Analysis; Mixed Model Analysis to evaluate interaction of group by time; Mean Difference (Final Values) = .04, Standard Error of Mean .029

5. Secondary Outcome: Overall Health- Short Form (36) Health Survey
Description: Short Form (36) Health Survey overall score ranges from 0 to 100. Computed as the mean of all SF-36 subscales.
  The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index. Lower scores are greater disability and higher scores are greater health functioning.
Time Frame: 6 months
Population: All participants who completed 1 or more SF-36 assessments were included in the analysis.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Physician Management | Physician Management Plus Cognitive Behavioral Therapy
Number analyzed (Participants) | 70 | 69
Scores on a scale | 75.3 (1.7) | 75.1 (1.6)
Statistical Analysis 1: Comparison: Physician Management vs Physician Management Plus Cognitive Behavioral Therapy; Test type: Superiority or Other; p = .24, Mixed Models Analysis; Mixed Model Analysis to evaluate interaction of group by time; Mean Difference (Final Values) = 2.38, Standard Error of Mean 3.63

ADVERSE EVENTS:
Arm/Group | Physician Management | Physician Management Plus Cognitive Behavioral Therapy
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/70
Other Adverse Events (participants affected / at risk) | 0/71 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No